CLINICAL TRIAL: NCT02680938
Title: Prophylactic Use of Intraumbilical Vein Oxytocin Injection in The Management of Third Stage of Labor A Randomized Controlled Study
Brief Title: Prophylactic Use of Intraumbilical Vein Oxytocin Injection in The Management of Third Stage of Labor
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, kareem Sami mostafa, lecturer assistant, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: gyn-057
Record Dates: First submitted 2016-02-04; First posted 2016-02-12 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2016-03

CONDITIONS: Postpartum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Oxytocin; Sodium Chloride

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- oxytocin group (Active Comparator): 10 units of oxytocin will be injected into the umbilical vein at the most proximal site to the placenta after clamping and cutting of the umbilical cord.
  Interventions: Drug: oxytocin
- control group (Placebo Comparator): 1 mL normal saline will be injected into the umbilical vein at the most proximal site to the placenta after clamping and cutting of the umbilical cord.
  Interventions: Drug: saline

INTERVENTIONS:
Drug: oxytocin — For each participant, the duration of the third stage of labor (the time period between the delivery of the fetus and the delivery of the placenta) will be recorded.
  - The two groups will be compared in the following terms:
  1. The duration of the third stage of labor by stopwatch.
  2. Hemoglobin (Hb) difference before and 12 h after delivery.
  3. The need for manual delivery of the placenta. Manual removal of the placenta will be commonly carried out under general sedation in the operating room, if the placenta will not be delivered 30 min after fetal delivery.
  Other Names: syntocinon
  Arms: oxytocin group
Drug: saline — For each participant, the duration of the third stage of labor (the time period between the delivery of the fetus and the delivery of the placenta) will be recorded.
  - The two groups will be compared in the following terms:
  1. The duration of the third stage of labor by stopwatch.
  2. Hemoglobin (Hb) difference before and 12 h after delivery.
  3. The need for manual delivery of the placenta. Manual removal of the placenta will be commonly carried out under general sedation in the operating room, if the placenta will not be delivered 30 min after fetal delivery.
  Other Names: placebo
  Arms: control group

SUMMARY:
The third stage is the interval between delivery of the infant and delivery of the placenta. This stage averages 10 minutes and is considered prolonged if it lasts longer than 30 minutes, placental separation occurs as a result of continued uterine contractions, continued contractions control blood loss by compression of spiral arteries and also result in migration of the placenta into the lower uterine segment and then through the cervix.

The intra-umbilical vein injection of 10 IU of oxytocin is recommended as a first line of treatment for retained placenta. Despite this recommendation, the method has yet to make its way into routine practice, probably because of the lack of a large substantive randomized controlled trial, and lingering doubts over which uterotonic to use and at what dosage.

The purpose of this study is to evaluate the effect of intraumbilical vein injection of oxytocin on reducing the duration of the third stage of labor and the need for manual delivery of placenta, ,in addition to reduce blood loss during third and fourth stage of labor and decrease incidence of rtained placenta in comparison with inraumblical injection of normal saline.

This is a prospective randomized control trial conducted at Ain Shams University Maternity Hospital. This study included 240 term pregnant women in labor admitted to the labor ward, They were divided into Two groups :

Group (A):

The experimental group, 10 units of oxytocin will be injected into the umbilical vein at the most proximal site to the placenta after clamping and cutting of the umbilical cord.

Group (B):

The control group, 1 mL normal saline will be injected into the umbilical vein at the most proximal site to the placenta after clamping and cutting of the umbilical cord.

DETAILED DESCRIPTION:
This study included 240 term pregnant women in labor admitted to the labor ward, They were divided into Two groups :

Group (A):

The experimental group, 10 units of oxytocin will be injected into the umbilical vein at the most proximal site to the placenta after clamping and cutting of the umbilical cord.

Group (B):

The control group, 1 mL normal saline will be injected into the umbilical vein at the most proximal site to the placenta after clamping and cutting of the umbilical cord.

complete blood count of both groups before and 12 h after delivery.

* The third stage of labor will be actively managed in the two groups by infusion of 20 IU oxytocin in 1 L Ringer's lactate solution at a rate of 100 mL/min, immediately after delivery of the fetus ( Nankali et al., 2013)..
* In the control group ( B ) , 1 mL normal saline will be injected into the umbilical vein at the most proximal site to the placenta after clamping and cutting of the umbilical cord.
* In the experimental group ( A ) , instead of normal saline, 10 IU (1mL) oxytocin will be injected at the same site. We will wait 30 min for the symptoms of placenta delivery (i.e., the uterus became firmer and more globular and was displaced upward, a gush of blood occurred, and the umbilical cord was elongated).
* Spontaneous delivery of the placenta will be achieved by touching the fundus and applying pressure on the symphysis pubis by a finger and slight traction of the umbilical cord.
* For each participant, the duration of the third stage of labor (the time period between the delivery of the fetus and the delivery of the placenta) will be recorded.
* The two groups will be compared in the following terms:

  1. The duration of the third stage of labor by stopwatch.
  2. Hemoglobin (Hb) difference before and 12 h after delivery.
  3. The need for manual delivery of the placenta. Manual removal of the placenta will be commonly carried out under general sedation in the operating room, if the placenta will not be delivered 30 min after fetal delivery.
  4. Estimate blood loss by Allowable Blood Loss (ABL) (Miller 2000)

ELIGIBILITY:
Inclusion Criteria:

1. 36 to 42 weeks gestational age.
2. Single alive fetus with cephalic presentation.
3. Parity 1 to 3.
4. Normal vaginal delivery.

Exclusion Criteria:

1. Placenta Previa.
2. Placental Abruption .
3. Prolonged Labor ( > 20 h )
4. History of Postpartum Hemorrhage or Antepartum Hemorrhage.
5. History of Cesarean delivery or any uterine scar .
6. Polyhydramnios .
7. Known uterine anomalies.
8. Coagulation disorders.
9. Abnormal placental adhesion.
10. Forceps or Vacuum delivery.
11. Chorioamninitis.
12. Multiple Gestations.
13. Accelerated Labor (< 3 h ).
14. Painless Labor with Epidural Anaethesia

Ages: 14 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Duration of the third stage of labor. | more than 30 minutes, we will do manual separation of placenta
  For each participant, the duration of the third stage of labor (the time period between the delivery of the fetus and the delivery of the placenta) will be recorded.

SECONDARY OUTCOMES:
Hb difference before and 12 h after delivery. | before labor and after 12 hours after delievery

CONTACTS AND LOCATIONS:
Overall Officials: kareem S mostafa, Principal Investigator — Ain Shams University
Locations (1):
- kareem Sami mostafa, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The aim of the present study was to evaluate the effect of intraumbilical vein oxytocin on reducing the duration of the third stage of labor and the need for manual delivery of placenta, in comparison with normal saline administration